CLINICAL TRIAL: NCT06521346
Title: The Effect of Active Cycle Breathing Technique on Respiratory Parameters, Dyspnea Related Kinesiophobia and Pain in Early Post Cardiac Surgery Patients
Brief Title: Active Cycle Breathing Technique (ACBT) on Respiratory Parameters, Dyspnea Related Kinesiophobia and Pain
Acronym: (ACBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Active cycle breath technique
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Complication; Cardiac Disease
Keywords: Respiratory function; Cardiac surgery
MeSH Terms: conditions — Heart Diseases; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: The total group will be divided into two group: control and intervention group Control group receives standard care in the unit Intervention group receives active cycle breathing techniques
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle breathing technique (Experimental): Breathing control phase Thoracic expansion exercises Forced expiration technique (huffing)
  Interventions: Procedure: Active cycle breathing technique
- Control group (Placebo Comparator): Patient who receives the routine care
  Interventions: Procedure: Routine care

INTERVENTIONS:
Procedure: Active cycle breathing technique — The ACBT was included if it was described as containing three essential components: 1) breathing control, 2) forced expiration technique and 3) thoracic expansion exercises. The technique may also include postural drainage (PD) or percussion/shaking.
  Arms: Active cycle breathing technique
Procedure: Routine care — Routine care delivers after extubating such as percussion or chest physiotherapy
  Arms: Control group

SUMMARY:
This study aims to improve pulmonary function impairment is associated with a reduction in chest expansion, lung volume, pain perception and an impairment of the Post cardiac surgery patient's ability to cough effectively. The technique of active cycle breathing consisted of three parts to the ACBT, which are:

* breathing control
* deep breaths
* huff or cough

DETAILED DESCRIPTION:
This study aims to explore the effect of Active Cycle Breathing Technique on Respiratory Parameters and Pain in Early Post Cardiac Surgery Patients

Research hypothesis:

-Post cardiac surgery patients who practice active breathing techniques exhibit an improvement in clinical outcomes compared to those who do not practice.

Research design:

A randomized control trial research design will be utilized to conduct this study.

Study Setting:

This study was carried out at the cardiac ICUs. A sample of 120 cardiac patients will be assigned in the current study from the previously mentioned settings.

The patients will be allocated into two equal groups, each with 60 patients. The control group will be composed of 60 patients who were managed by routine cardiac care The study group will consist of 60 patients who were exposed to an active cycle of breathing techniques

Inclusion criteria:

* Adult patients of both genders.
* After extubating for at least 6 hours
* Hemodynamic stable patients
* Able to communicate. Exclusion criteria: Patient with complication postoperative surgery Patient's demographic characteristics as patient's code, age, gender, marital status, education, and occupation.

Study group: managed by the use of active cycle breathing techniques combined with routine physiotherapy.

* Each session of the active cycle breathing technique lasted for 10 to 20 minutes.
* The active cycle breathing technique was carried out for three days post extubating four sessions done daily.

Implementation of active cycle breathing technique

* Explain the steps of ACBT to the patient.
* The patient was placed in a semi-sitting position with her or his back straight, and instructions were given to the patient to do the following steps:

  1 . Breathing control phase
* Hold the spirometer straight.
* Exhale, then seal your lips around the mouthpiece and inhale slowly and deeply into your mouth.
* The piston in the incentive spirometer's transparent chamber will rise when you inhale deeply.
* Hold your breath for 3 to 5 seconds after taking a deep breath.
* Remove the mouthpiece and slowly exhale. For a few seconds, until the piston descends to the bottom of the chamber, relax and breathe normally.
* To regain control of their breathing, the patient was told to do lengthy, slow expirations between 5 and 7 times.

  2 . Thoracic expansion exercises The patient was instructed to relax your upper chest.
* The patient was instructed to breathe slowly and deeply through the nose without using the accessory muscle.
* The patient was instructed to hold their breath initially for 3 to 4 seconds and gradually increase it to the maximum time.

Don't force the breath out; instead, softly exhale through pursed lips until your lungs are empty.

* Repeat the previous steps from 3to4 times. 3- Forced expiration technique (huffing)
* Patient was instructed to support the incision site by using a chest binder or keeping your hands over your incision.
* Cough twice as many times as they huffed two to three times.
* This step was repeated a minimum of two times and a maximum of three times in one session.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders.
* After extubating for at least 6 hours post operation.
* Hemodynamic stable patients
* Able to communicate.

Exclusion Criteria:

* Instability of patient's medical condition or hemodynamic instability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Respiratory parameters | Three observation days
  change in respiratory rate
Pain perception | Three observation days
  Using visual analogue scale score 0 mean no pain while score 10 means sever pain
Dyspnea-related kinesiophobia | preoperative, three observation days, and day of discharge
  comprises 11 items include five items dyspnea and six items for fear of activity dimension and each item is rated from "strongly disagree" (score = 1) to "strongly agree" (score = 5) for a total score between 11 and 55.

SECONDARY OUTCOMES:
Deterioration in clinical parameters such as vital signs | Three observation days
  hypoxic event
ICU and hospital stay | three observation days
  ICU and hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of nursing Damanhour university, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewis LK, Williams MT, Olds TS. The active cycle of breathing technique: a systematic review and meta-analysis. Respir Med. 2012 Feb;106(2):155-72. doi: 10.1016/j.rmed.2011.10.014. Epub 2011 Nov 18. PMID 22100537
- [Background] Mckoy NA, Wilson LM, Saldanha IJ, Odelola OA, Robinson KA. Active cycle of breathing technique for cystic fibrosis. Cochrane Database Syst Rev. 2016 Jul 5;7(7):CD007862. doi: 10.1002/14651858.CD007862.pub4. PMID 27378490